CLINICAL TRIAL: NCT03748550
Title: EXercise to Prevent AnthraCycline-based Cardio-Toxicity 2.0 (EXACT2) in Individuals With Breast Cancer
Brief Title: Exercise to Prevent AnthraCycline-based Cardio-Toxicity Study 2.0 (EXACT2)
Acronym: EXACT2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1024489; 1024489 (Other: Nova Scotia Health Authority)
Record Dates: First submitted 2018-11-13; First posted 2018-11-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cancer, Breast; Cardiotoxicity; Cardiovascular Diseases
Keywords: Anthracyclines; Cardiotoxic; Breast cancer; Aerobic exercise; Cardiac structure; Cardiac function; CVD risk
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either the standard of care group (control) or the intervention group (standard of care + 12-weeks aerobic exercise).
Who Masked: Outcomes Assessor
Masking Description: Clinicians interpreting the echocardiograms and stress test results will not know whether the participant is in the control group or the exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive standard of care treatment for their breast cancer.
- Exercise (Experimental): Participants will receive standard of care treatment for their breast cancer plus be given a 12-week home based aerobic exercise program.
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — All participants will receive standard of care for their cancer as well as given a 12-week, home-based progressive aerobic exercise (AE) program. A nonlinear progressive training approach will be used whereby each participant will perform two AE sessions (e.g. walking), on non-consecutive days, per week. AE sessions will vary between low (35-45% heart rate reserve (HRR)), low-moderate (46-55% HRR), high-moderate (56-70% HRR) and high (71-85% HRR) intensity.
  Arms: Exercise

SUMMARY:
Although great progress has been made in treating breast cancer, long-term health may be impaired by cancer therapy. For example, some chemotherapy drugs (e.g., anthracyclines) are known to cause declines in heart health. While the impact can vary, some will experience substantial heart damage that may lead to heart failure and death. As these treatments are highly effective, there is a need to find ways to reduce the damaging effects while not interfering with its anticancer potential. As it is well-known that regular exercise can improve heart health, the purpose of this study is to explore the role of exercise as a heart protective therapy for breast cancer patients receiving heart damaging chemotherapy.

DETAILED DESCRIPTION:
As a result of advances in cancer treatment, the number of breast cancer (BC) survivors is increasing in Canada. Unfortunately, the drugs used to treat BC can have a negative impact on the long term health and welfare of the BC survivors (BCS). For example, commonly used cancer therapies, such as anthracyclines (AC) are known to cause declines in heart health. While the impact can vary, some individuals treated with these medications will experience substantial heart damage that may lead to heart failure and death. As a result, risk of cardiovascular morbidity/mortality has become a major concern for BCS that received AC treatment. As a result, there is an immediate need to find therapies that can be used to prevent damage to the heart without limiting the anticancer potential of AC.

A growing body of evidence suggests that aerobic exercise training may help protect the heart against the damaging effects of AC therapy. These studies, which were conducted using animal models, have shown that performing aerobic exercise before or while undergoing AC therapy helps to maintain heart function and prevent structural changes in the heart. However, to the author's knowledge similar studies have not been conducted in BCS undergoing treatment, thus it remains unclear whether exercise has the same cardioprotective effect in BCS. As a first step in answering this question, our research group conducted a pilot study that showed a 12-week aerobic exercise program is safe and feasible for BCS undergoing chemotherapy. The next step in our research is to determine whether aerobic exercise decreases or prevents cardiotoxicity in BCS receiving AC treatment. Therefore, the purpose of this study is to determine whether a 12-week home based aerobic exercise program mitigates AC-mediated cardiotoxicity in BCS on active treatment. The specific objectives of the study are to determine whether the aerobic exercise program: 1) prevents structural and functional changes in the heart; 2) maintains peak aerobic capacity throughout the treatment process; and 3) decreases biological markers associated with heart damage.

This is a randomized control trial with repeated measures. BCSs will be randomly assigned to either the wait-list control (CTL) group (standard of care (SOC) or the aerobic exercise (AEX; SOC + 12-week home-based aerobic exercise program). One hundred BCS (18-65 years of age) on AC treatment will be recruited from two sites, Halifax, NS (n=50) and Winnipeg, MB (n=50). Patients in the AEX group will perform two exercise sessions per week that will range from low intensity (~45 min) to vigorous intensity (~20 min). BCS will monitor their exercise intensity with Polar A370 HR monitors, which they will be given for the duration of the study.The primary outcome measure for the study is cardiac function as determined by echocardiography and a cardiac stress test. Secondary outcome measures include serum biomarkers associated with cardiotoxicity (e.g. c-reactive protein, hsTNT, NT-proBNP). Patient-reported outcomes including levels of fatigue and quality of life will also be assessed. The study outcome measures will be assessed prior to the participants starting AC therapy (week-0), post-exercise intervention (week-12) and 6 months after the completion of the AEX. Of note, upon completion of the 6 month follow-up testing participants in the CTL group, if interested, will be given the home-based AEX as well the necessary support to complete the program.

This research will provide the first direct evidence that aerobic exercise protects the heart from AC-mediated damage in BCS undergoing cancer treatment. Both the medical and research communities will benefit from this research as it could lead to the improvement of long term health of cancer survivorship as well as improve the understanding of how the heart health can be maintained during cancer therapy. Given the significant impact of AC therapy on improving BC prognosis, and the potential protective effects of exercise training, this study will be important in improving BC care via the improvement of the quality of life and increased survivorship.

ELIGIBILITY:
Inclusion Criteria:

* 1) must be 18 years or older.
* diagnosed with breast cancer (stages I-III) and not have started therapy.
* must be scheduled to receive AC- based chemotherapy (minimum dose of 240 mg/m2 of DOX or 300 mg/m2 of DAN).
* are able to undertake a 12-week home-based, progressive aerobic exercise program.
* have medical clearance from a cardiologist (e.g. based on stress test results) to participate in the study.

Exclusion Criteria:

* significant cognitive limitations.
* pre-existing medical condition that would otherwise contraindicate aerobic exercise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular (LV) Function | LV function will be assessed at baseline (week 0), post-intervention (week-13) and 6 months after the completion of the intervention.
  LV function will be assessed using serial transthoracic echocardiography (TTE) as well as tissue velocity imaging (TVI) and strain imaging (SI.) For 2-dimensional (2D) LV cavity dimensions and LVEF will be determined from the acquired 2D images according to established criteria. Tissue Doppler-derived indexes will be recorded at the base of the lateral mitral annuli to determine longitudinal endocardial velocities. The indexes that will be assessed are systolic (S'), early diastolic (e') and late diastolic (a') velocities. Doppler-independent strain will be assessed offline using semi-automated speckle tracking techniques. These will be performed using parasternal and apical views to determine both global longitudinal and radial strain.

SECONDARY OUTCOMES:
Change in Cardiac Electrical Activity | The cardiac ECG will be assessed at baseline (week 0), post-intervention (week-13) and 6 months after the completion of the intervention.
  Cardiac electrocardiogram at rest will be assessed using a 12 lead ECG (General Electric Case System). Specifically, the duration (ms) of the PR interval, RR interval, QRS interval and QT interval will be determined.
Change in Aerobic Fitness | Outcome will be assessed at baseline (week 0), post-intervention (week-13) and 6 months after the completion of the intervention.
  Cardiac Stress Tests results will be used to predict peak oxygen consumption (ml/kg/min). In brief, participants will perform a graded exercise test until they reach volitional fatigue or the test is terminated due to adverse physiological changes. Predictive equations will then be used to predict the participant's peak oxygen uptake based on the total duration (seconds) of the treadmill test.
Change in Blood biomarkers | Outcome will be assessed at baseline (week 0), post-intervention (week-13) and 6 months after the completion of the intervention.
  Venipuncture will be performed by a nurse/phlebotomist to collect blood samples which will be used to quantify systemic levels of c-reactive protein (CRP), high sensitivity troponin (hs-TNT) and NTproBNP levels. Upon collection, blood samples will be processed, and the serum will be extracted and stored at -20°C until it is required for analysis. CRP, hs-TNT and N-terminal pro b-type natriuretic peptide (NTproBNP) levels will be assessed using commercially available ELISA kits. All biomarkers will be measured in pg/ml.
Change in Functional Assessment for Cancer Therapy | Outcome will be assessed at baseline (week 0), post-intervention (week-13) and 6 months after the completion of the intervention.
  The Functional Assessment for Cancer Therapy survey for patients with breast cancer (FACT-B) will be used to assess quality of life. The FACT-B includes sub-scales for assessing physical, social/family, emotional, and functional well-being. FACT-B total score ranges from 0-148.
Change in Fatigue | Outcome will be assessed at baseline (week 0), post-intervention (week-13) and 6 months after the completion of the intervention.
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) is a 13 item questionnaire (maximum score =160) that will be used to assess cancer-related fatigue. Higher scores are indicative of higher levels of fatigue.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No